CLINICAL TRIAL: NCT02902744
Title: Fluocinolone Acetonide Insert (ILUVIEN®) for Diabetic Macular Edema (FAD) Study
Acronym: FAD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was withdrawn due to difficult recruitment of patients for the study; No participants were enrolled in the study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00082826
Record Dates: First submitted 2016-09-12; First posted 2016-09-16 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Fluocinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ILUVIEN 0.19 MG (Experimental)
  Interventions: Drug: ILUVIEN®

INTERVENTIONS:
Drug: ILUVIEN® — Patients will receive Iluvien as the standard of care treatment for diabetic macular edema.
  Other Names: Fluocinolone Acetonide Intravitreal Implant 0.19 mg

SUMMARY:
Primary Objective:

• To collect post-approval safety data related to intraocular pressure (IOP) after one or more injections of Iluvien as standard of care in subjects with diabetic macular edema (DME).

Secondary Objectives:

• To collect visual and anatomic outcome data after one or more injections of Iluvien as standard of care in subjects with diabetic macular edema (DME).

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is a major complication of diabetes mellitus that can lead to significant visual morbidity. Important features of DR are microaneurysms, vascular leakage, vascular occlusion, and retinal neovascularization. Diabetic macular edema (DME) occurs when there is leakage in the macula, the central region of the retina that is responsible for fine visual acuity. DME is the most prevalent cause of moderate visual loss in patients with diabetes.(1)

Treatment options for DME include the use of focal/grid laser photocoagulation (2), intravitreal anti-VEGF therapy (3-5), intravitreal steroid therapy (6) and steroid implant insertion into the vitreous cavity (7-9).

Corticosteroids are known to be beneficial in the treatment of DME by reducing the expression of vascular endothelial growth factor (VEGF) and other inflammatory cytokines e.g. Interleukin-6, which play a major role in pathogenesis of DME. (10).

Iluvien® (Alimera Sciences, Inc., Alpharetta, GA) is a low dose, sustained release corticosteroid insert that has recently been FDA approved for use in patients with DME. (10, 11) Structurally it is a nonbiodegradable, cylindrical polymer tube measuring 3.5x0.37 mm which releases 0.19 µg/day of Fluocinolone Acetonide. These inserts are injected into the vitreous cavity in an outpatient setting through a 25-gauge injector system which uses MedidurTM (Alimera Sciences, Inc.) technology and are found to be beneficial compared to sham treatment for up to 3 years. (10, 11) As a complication steroid implants can sometimes result in a dose dependent elevation in the intraocular pressure (IOP) which can increase the risk of glaucoma in susceptible patients. The purpose of this study is to look at post-approval safety data related to IOP after one or more injections of Iluvien as standard of care in subjects with DME.

Objectives

Primary Objective:

• To collect post-approval safety data related to intraocular pressure (IOP) after one or more injections of Iluvien as standard of care in subjects with diabetic macular edema (DME).

Secondary Objectives:

• To collect visual and anatomic outcome data after one or more injections of Iluvien as standard of care in subjects with diabetic macular edema (DME).

Study Procedures

This study will assess the long term safety, visual, and anatomic outcomes in subjects receiving 1 or more injections of Iluvien as standard care for DME. Fifty patients from the clinic population of the Wilmer Eye Institute will be enrolled in the study for a duration of 60 months. Subjects will have a measurement of best corrected visual acuity (BCVA), IOP and eye exam at baseline and months 12, 24, 36, 48, and 60. All other follow up and all treatment will be in the clinic by the patient's treating physician. Data from the clinic notes will be collected on case report forms and adverse events will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Subjects receiving Iluvien as standard of care for DME
* Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure.

Exclusion Criteria:

• None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Percentage of patients that require a surgical procedure for increased IOP that could not be controlled by IOP-lowering drops. | 5 years
  Percentage of patients that require a surgical procedure for increased intraocular pressure that could not be controlled by IOP-lowering drops.
Percentage of patients requiring 1, 2, or 3 medications to control IOP. | 5 years
  Percentage of patients requiring 1, 2, or 3 medications to control intraocular pressure.
Percentage of patients with IOP > 25mmHg on two occasions and percentage of patients with IOP > 30mmHg on two occasions | 5 years
  Percentage of patients with intraocular pressure > 25mmHg on two occasions and percentage of patients with intraocular pressure > 30mmHg on two occasions
Percentage of patients losing > 15 letters at month 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60 | 5 years
  Percentage of patients losing > 15 letters at month 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60

SECONDARY OUTCOMES:
Mean change from baseline BCVA ETDRS letter score at months 12, 24, 36, 48, and 60 | 5 years
  Mean change from baseline best corrected visual acuity (BCVA) ETDRS letter score at months 12, 24, 36, 48, and 60
Mean change from baseline CST measured by spectral domain-optical coherence tomography (SD-OCT) at months 12, 24, 36, 48, and 60 | 5 years
  Mean change from baseline central subfield thickness (CST) measured by spectral domain-optical coherence tomography (SD-OCT) at months 12, 24, 36, 48, and 60
Percentage of subjects with gain from baseline BCVA letter score ≥ 15; ≥ 10; ≥ 5 at months 12, 24, 36, 48, and 60 | 5 years
  Percentage of subjects with gain from baseline best corrected visual acuity (BCVA) letter score ≥ 15; ≥ 10; ≥ 5 at months 12, 24, 36, 48, and 60
Percentage of subjects with CST ≤300µm at months 12, 24, 36, 48, and 60 | 5 years
  Percentage of subjects with central subfield thickness (CST) ≤300µm at months 12, 24, 36, 48, and 60
Percentage of subjects with no intraretinal or subretinal fluid in the macula at months 12, 24, 36, 48, and 60 | 5 years
  Percentage of subjects with no intraretinal or subretinal fluid in the macula at months 12, 24, 36, 48, and 60
Number of anti-VEGF injections required between baseline and month 60 | 5 years
  Number of anti-VEGF injections required between baseline and month 60

CONTACTS AND LOCATIONS:
Overall Officials: Gulnar Hafiz, MD, MPH, Study Director — Wilmer Eye Institute, Johns Hopkins Hospital
Locations (1):
- Wilmer Eye Institute, Johns Hopkins University School of Medicine, Baltimore, Maryland, United States